CLINICAL TRIAL: NCT04983680
Title: Remote-delivered Mindfulness-Based Cognitive Therapy to Target Fear of Recurrence Among SCAD Survivors
Brief Title: Remote-delivered MBCT for SCAD Survivors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christina Luberto, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P001519; P30AG064198 (NIH)
Record Dates: First submitted 2021-07-13; First posted 2021-07-30 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease; Anxiety; Sleep
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-Based Cognitive Therapy (Experimental): Mindfulness-Based Cognitive Therapy (MBCT) is an 8-week group intervention (1.5-hour weekly sessions) that combines cognitive-behavioral therapy and mindfulness training to treat emotional problems.
  Interventions: Behavioral: MBCT

INTERVENTIONS:
Behavioral: MBCT — Mindfulness-Based Cognitive Therapy (MBCT) is an 8-week group intervention (1.5-hour weekly sessions) that combines cognitive-behavioral therapy and mindfulness training. In this study, MBCT has been adapted to include education about cardiac health and fear of recurrence, and the intervention is delivered remotely via synchronous group videoconference. There is 15-20 minutes of daily mindfulness practice between sessions. Participants are provided a home practice record form and asked to submit the completed form to study staff each week.

SUMMARY:
Spontaneous coronary artery dissection (SCAD) is an important cause of cardiac events, primarily affecting young healthy women with no cardiovascular risk factors. The 10-year recurrence rate is 30%, but SCAD recurrence cannot be predicted. Approximately half of SCAD survivors struggle with significant anxiety and fear of recurrence (FOR), which contributes to poor sleep and physical inactivity and, thereby, increased risk of recurrence. Mindfulness-Based Cognitive Therapy (MBCT) is an 8-week group intervention with evidence to improve FOR and health behaviors (sleep, physical activity), through psychological mechanisms that directly target key FOR processes (interoceptive bias, intolerance of uncertainty). I adapted MBCT to target FOR, sleep, and physical activity in cardiac event survivors via group videoconferencing delivery (UpBeat-MBCT), however this intervention has not yet been targeted to SCAD survivors. I propose an open pilot trial to test the feasibility, acceptability, and changes in psychological and behavioral health variables in SCAD survivors participating in UpBeat-MBCT (N=16). Participants will be recruited from the MGH SCAD Program and asked to complete self-report surveys and actigraphy before and after the intervention. The primary outcomes are feasibility and acceptability of the intervention and research procedures. Exploratory outcomes are changes in psychological and behavioral variables and their inter-correlations. This project would be the first and only behavioral intervention for SCAD survivors and would provide preliminary data for an NIH Stage II efficacy trial to develop an accessible and efficacious intervention for a vulnerable group of SCAD survivors, with generalizability to survivors of other cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Cardiologist-confirmed diagnosis of SCAD in the past 1-12 months
* English-speaking and reading
* Internet access (via computer or mobile device).

Exclusion Criteria:

* Terminal illness with life expectancy <1 year
* Severe mental illness requiring urgent psychiatric intervention (e.g., active suicidal ideation) or past-year psychiatric hospitalization)
* Significant cognitive impairment preventing informed consent determined by study staff or medical record review (e.g., medical history of cognitive impairment)
* Deemed unable to complete research procedures (e.g., group sessions or surveys) per clinical judgment of study staff
* Unavailable for intervention sessions (e.g., schedule conflicts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Luberto, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mongan Institute: Health Policy Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luberto CM, Lopes M, Cloutier JG, Hall DL, Wood M, Schuman-Olivier Z, Hoeppner BB, Park ER. Remotely delivered mindfulness-based cognitive therapy for spontaneous coronary artery dissection survivors. Transl Behav Med. 2025 Jan 16;15(1):ibaf064. doi: 10.1093/tbm/ibaf064. PMID 41120129

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-Based Cognitive Therapy
Started | 19
Completed | 12
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.68 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis population for gender is n=17 which differs from the overall sample (n=19) because two participants did not report their gender.
  Participants
    number analyzed (Participants) | 17
    Female | 16
    Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Time Since SCAD [Mean (Standard Deviation); unit: months] | 22.74 (4.24)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrollment: Percent of Participants Enrolled
Description: Feasibility will be assessed by >70% of eligible patients enroll
Time Frame: 7 months
Population: The number of participants analyzed for this variable (n=20) is higher than the number who started the trial (n=19), because one person who screened eligible refused to enroll.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 20
Participants | 19

2. Primary Outcome: Feasibility of Retention: Percent of Enrolled Participants Retained at Post-intervention
Description: Feasibility of retention will be assessed by > 70% of participants completing the post-intervention survey
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 19
Participants | 12

3. Primary Outcome: Feasibility of Daily Diaries: Percent of Participants Who Complete the Daily Diaries at Pre-intervention
Description: Feasibility of daily diary completion will be assessed by >70% of participants completing daily diaries for 7 consecutive days at pre-intervention
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 19
Participants | 13

4. Primary Outcome: Feasibility of Daily Diaries: Percent of Participants Who Complete the Daily Diaries at Post-intervention
Description: Feasibility of daily diary completion will be assessed by >70% of participants completing daily diaries for 7 consecutive days at post-intervention
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
Participants | 7

5. Primary Outcome: Feasibility of Actigraphy Use: Percent of Participants Who Adhere to Actigraphy Procedures at Pre-intervention
Description: Feasibility of actigraphy use will be assessed by >70% of participants completing actigraphy for 7 consecutive days at pre-intervention
Time Frame: 7 months
Population: Participants who received an actigraphy watch as part of the study. Note that although 19 participants were enrolled, only 18 received a watch and were included in actigraphy procedures because the study team only had 18 watches available.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 18
Participants | 18

6. Primary Outcome: Feasibility of Actigraphy Use: Percent of Participants Who Adhere to Actigraphy Procedures at Post-intervention
Description: Feasibility of actigraphy use will be assessed by >70% of participants completing actigraphy for 7 consecutive days at post-intervention
Time Frame: 7 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 18
Participants | 13

7. Primary Outcome: Feasibility of MBCT Intervention: Participant Attendance Rates
Description: Feasibility of UpBeat-MBCT intervention will be assessed by >70% of participants attending >6/8 sessions
Time Frame: 7 months
Population: participants who enrolled in, and attended, group intervention sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 19
Participants | 10

8. Primary Outcome: Feasibility of Videoconferencing Delivery: Percent of Sessions With Videoconferencing Problems
Description: Feasibility of videoconferencing delivery will be assessed by <20% of sessions missed due to videoconference problems
Time Frame: 7 months
Measure: Count of Units; unit: Number of virtual sessions
Units Other Than Participants: Number of virtual sessions
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 19
Number analyzed (Number of virtual sessions) | 16
Number of virtual sessions | 0

9. Primary Outcome: Intervention Acceptability: Plans to Use the Skills in the Future
Description: Intervention acceptability will be assessed by >70% plan to use the intervention skills in the future
Time Frame: 7 months
Population: Participants retained at post-intervention who answered this item on the post-survey
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 11
Participants | 11

10. Primary Outcome: Intervention Acceptability: Would Recommend the Program to Others
Description: Intervention acceptability will be assessed by >70% would recommend the program to others
Time Frame: 7 months
Population: Participants retained at post-intervention who answered this item on the post-survey
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 11
Participants | 10

11. Primary Outcome: Intervention Acceptability: Home Practice Completion
Description: Acceptability of the UpBeat-MBCT intervention will be assessed by >70% of participants completing home practice >3days/week
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
Participants | 9

12. Primary Outcome: Acceptability of Daily Diary Surveys: Ease of Completion
Description: Acceptability of daily diaries will be assessed by ease of daily diary completion (1=not at all, 10=extremely). Mean acceptability rating > 7.0 indicates acceptability
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
score on a scale | 7.83 (2.21)

13. Primary Outcome: Acceptability of Daily Diary Surveys: Level of Survey Interference
Description: Acceptability of daily diaries will be assessed by level of survey interference in daily life (1=not at all, 10=extremely, M<2.0)
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
score on a scale | 3.0 (2.59)

14. Primary Outcome: Acceptability of Actigraphy
Description: Acceptability of actigraphy will be assessed by ratings of ease of actigraphy completion (1=not at all, 10 =extremely, M>7.0)
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
score on a scale | 8.67 (2.27)

15. Secondary Outcome: Fear of Recurrence
Description: The Assessment of Survivor Concerns, a validated self-report survey, will be used to explore the severity of fears of recurrent cardiac events before and after the intervention. This study used a 5 item version of the ASC, thus the scores range from 5 (lower fear of reoccurrence) to 20 (higher fear of reoccurrence). The 5 item version has two subscales: health worry, cardiac worry. Scores from each subscale are summed to achieve the final score.
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
score on a scale
  Pre-intervention | 13.33 (3.50)
  Post-intervention | 11.33 (3.85)

16. Secondary Outcome: Cognitive De-centering
Description: The Experiences Questionnaire, a validated self-report survey, will be used to explore levels of trait cognitive de-centering before and after the intervention (i.e., the ability to notice mental events as transient objects separate from the self). Each item is scored on a Likert scale from 1 (never) to 5 (all of the time); the total minimum score is 11 while the maximum score is 55. Higher scores indicate greater cognitive decentering (better outcomes), while lower scores indicate less cognitive de-centering (worse outcome)
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 11
score on a scale
  Pre-intervention | 32.91 (10.00)
  Post-intervention | 38.18 (6.52)

17. Secondary Outcome: Distress Tolerance
Description: The Distress Tolerance Scale, a validated self-report survey, will be used to explore levels of the ability to withstand negative emotional states before and after the intervention. The DTS is 15 item measure where each item is scores from 1 (strongly agree) to 5 (strongly disagree). Lower scores (minimum = 1) indicate lower distress tolerance and worse outcomes. Higher scores (maximum = 5) indicate higher distress tolerance and better outcomes.
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 11
score on a scale
  Pre-intervention | 3.19 (.94)
  Post-intervention | 3.39 (.76)

18. Secondary Outcome: Attention Regulation
Description: The Cognitive Affective Mindfulness Scale-Revised, a validated self-report survey, will be used to explore levels of trait mindfulness before and after the intervention. Items are scored on a scale 1 (Rarely/Not at all) to 4 (Almost Always). Lower scores (minimum = 1) reflect lower trait mindfulness (worse outcome) whereas higher scores (maximum = 40) indicate higher trait mindfulness (better outcome)
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
score on a scale
  Pre-intervention | 31.58 (8.74)
  Post-intervention | 32.58 (6.93)

19. Secondary Outcome: Non-judgmental Body Awareness
Description: The body trusting subscale of the multidimensional assessment of interoceptive awareness, a validated self-report survey, will be used to explore levels of non-judgmental body awareness before and after the intervention. The minimum score on the subscale is 0 while the maximum is 10. Scores of 10 indicate higher body trusting (better outcome). Scores of 0 indicate lower body trusting (worse outcome).
Time Frame: 7 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 8.0 (5.54)
  Post-intervention | 8.7 (4.76)

20. Secondary Outcome: Interoceptive Bias
Description: The Body Vigilance Scale, a validated self-report survey, will be used to explore attentional bias, hypervigilance, and sensitivity toward physical sensations around the chest before and after the intervention. The maximum score is 280, indicating high body vigilance and worse outcomes, while the minimum score is 0,indicating low body vigilance and better outcomes.
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
score on a scale
  Pre-intervention | 18.25 (5.28)
  Post-intervention | 15.08 (5.14)

21. Secondary Outcome: Intolerance of Uncertainty
Description: The Intolerance of Uncertainty Scale-12, a validated self-report survey, will be used to explore the ability to tolerate uncertainty before and after the intervention. The maximum score is 60 which indicates high intolerance of uncertainty and worse outcomes. The minimum score is 12 which indicates low intolerance of uncertainty and better outcomes. Each item is scored on a scale from 1 (not at all characteristic of me) to 5 (entirely characteristic of me).
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 11
score on a scale
  Pre-intervention | 33.36 (14.40)
  Post-intervention | 27.63 (12.91)

22. Secondary Outcome: Cardiac Anxiety
Description: Four items from the physical concerns subscale of the Anxiety Sensitivity Index 3 will be used to assess cardiac anxiety levels before and after the intervention. Items are scored on a scale from 0 (very little) to 4 (very much). The minimum possible score is 0, indicating low anxiety sensitivity and better outcomes. The maximum possible score is 16, indicating high anxiety sensitivity and worse outcomes.
Time Frame: 7 months
Population: N=8 in post intervention due to incomplete surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
score on a scale
  Pre-intervention | 9.42 (4.21)
  Post-intervention: number analyzed (Participants) | 8
  Post-intervention | 6.83 (4.61)

23. Secondary Outcome: Self-reported Sleep Outcomes
Description: Sleep duration, sleep efficiency, and sleep onset latency will be assessed by self-report survey via the Consensus Sleep Diary before and after the intervention and will be included in the sleep diaries.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: number of awakenings per night
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
number of awakenings per night
  Pre-Intervention | 1.83 (1.11)
  Post-Intervention | 1.63 (0.92)

24. Secondary Outcome: Self-reported Physical Activity
Description: Moderate-vigorous physical activity engagement will be assessed by self-report survey via the Physical Activity Vital sign before and after the intervention, including daily diaries.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: hours/week
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 12
hours/week
  Pre-Intervention | 33.46 (27.11)
  Post-Intervention | 59.50 (55.45)

ADVERSE EVENTS:
Time Frame: The data were collected over 7 months.
Arm/Group | Mindfulness-Based Cognitive Therapy
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness-Based Cognitive Therapy (N=19)
Adverse Event (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT04983680/Prot_SAP_000.pdf